CLINICAL TRIAL: NCT05909371
Title: Physiotherapy and Rehabilitation Doctoral Thesis Work
Brief Title: Investigation of the Effects of Motor Cognitive Dual Task Exercises on Cognitive Function, Balance and Functional Capacity in Patients Who Have Undergone Liver Transplantation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, İlker DEMİR, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Hasankalyoncüüniversityilker
Record Dates: First submitted 2023-05-22; First posted 2023-06-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical physiotheraphy (Experimental): The Program Applied to the Classical Physiotherapy Group The Warm-Up The postural exercises Short Breathing exercises Strengthening exercises Don't sit up Daily Balance exercises Walking exercises Pre-cooling exercise An individual-specific standardized exercise program suitable for clinical characteristics will be applied to patients with a maximum of 1 set of 8-12 repetitions for 30-45 minutes for each exercise (Modified Borg scale 4-6).
  Interventions: Other: exercise
- Motor cognitive exercise group (Experimental): The Program to be Applied in addition to the Physiotherapy Program to the Motor-cognitive Exercise Group .Remembering the word. Color/week/month/animal names counting/// girls boy names counting/// Country City names counting.
  from 50 back to 2 bad, 3 er,// counting from 50 back to 4 er//counting from 100 back to 2 bad 2 bad 3 er 3 er and simple arithmetic problems with single digits.
  Counting the months of the year// Counting the months of the year starting from any month// Counting the months of the year and 30 31 days.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Application of two different exercises to liver transplant individuals.

SUMMARY:
Liver transplantation is a life-saving treatment of choice for patients with acute or chronic liver failure. Liver transplantation is performed with a graft taken from a living donor or cadaver in patients with end-stage liver failure or who develop various complications regardless of the stage of the disease.In liver diseases, cognitive problems occur as well as physical problems. It has been observed that in some liver diseases, including hepatitis C, Wilson's disease, primary biliary cirrhosis, cognitive dysfunction that negatively affects the quality of life of patients, from mild cognitive problems to hepatic encephalopathy.

Our study will be carried out in Malatya İnönü University Turgut Özal Medical Center Liver Transplant Institute Hospital in order to investigate the effects of motor-cognitive dual-task exercises on cognitive function, balance and functional capacity in liver transplant patients.It will be divided into 2 groups as classical physiotherapy and motor-cognitive exercise. Classical physiotherapy and motor-cognitive exercise programs will be applied to the groups in accordance with the clinical characteristics of the individuals, tolerable, and in a standardized manner specific to the individuals. Evaluations will be made on the first day and at the end of the twenty-fourth session while the patient is in the service before starting the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be able to mobilize alone
* Having performed a liver transplant over the age of 50
* Spontaneous breathing
* Being hemodynamically stable
* Ability to read and write
* Not having an orthopedic disability and functional capacity limitation
* Being conscious and cooperative

Exclusion Criteria:

* Not agreeing to participate in the study
* Not continuing the treatment regularly
* Having neurological or neuropsychiatric problems
* Being colorblind

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Cognitive Functions | One day
  The Montreal Cognitive Assessment Scale will be used to evaluate cognitive functions. The score is between 0-30 points. In order to be considered as a cognitive disorder, the participant must get a score below 21 points.
Evaluation of Cognitive Functions | One day before the rehabilitation
  The Montreal Cognitive Assessment Scale will be used to evaluate cognitive functions. The score is between 0-30 points. In order to be considered as a cognitive disorder, the participant must get a score below 21 points. A day before the rehabilitation
Evaluation of Balance | One day before the rehabilitation
  Functional reach and timed get-go test were used for dynamic balance assessment, and single-leg standing tests were used for static balance assessment. A day before the rehabilitation
Evaluation of Balance | One day
  Functional reach and timed get-go test were used for dynamic balance assessment, and single-leg standing tests were used for static balance assessment.At the time of discharge
Assessment of functional capacity | One day before the rehabilitation
  In order to determine the functional capacity, a 6-minute walking test was applied. A day before the rehabilitation
Assessment of functional capacity | One day
  In order to determine the functional capacity, a 6-minute walking test was applied.At the time of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)